CLINICAL TRIAL: NCT02947204
Title: Intermittent vs. Continuous Oxygen Saturation Monitoring in Infants Hospitalized for Bronchiolitis: A Randomized Controlled Trial
Brief Title: Oxygen Saturation Monitoring in Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Sanjay Mahant, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1000054699
Record Dates: First submitted 2016-10-20; First posted 2016-10-27 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Length of Hospital Stay; Clinical Trial; Oxygen Saturation Monitoring
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous oxygen monitoring (Active Comparator): Oxygen saturation will be measured continuously through the child's hospital stay until discharge.
  Interventions: Other: Continuous oxygen monitoring
- Intermittent oxygen monitoring (Experimental): Oxygen saturation will be measured intermittently, every 4 hours, through the child's hospital stay until discharge.
  Interventions: Other: Intermittent oxygen monitoring

INTERVENTIONS:
Other: Intermittent oxygen monitoring — Oxygen saturation and vital signs will be measured intermittently at a frequency of every 4 hours by the bedside nurse through the child's hospital stay until discharge. Vital signs will be completed every 4 hours.
  Other Names: Intermittent
  Arms: Intermittent oxygen monitoring
Other: Continuous oxygen monitoring — Oxygen saturation will be measured continuously through the child's hospital stay until discharge. Vital signs will be completed every 4 hours.
  Other Names: Continuous
  Arms: Continuous oxygen monitoring

SUMMARY:
The investigators will conduct a study around the best way to monitor infants hospitalized with bronchiolitis, the most common lung infection and a leading reason for hospitalization in infants. Infants with bronchiolitis have breathing difficulties and are provided supplemental oxygen if their oxygen levels are low. However, there is uncertainty regarding how to best monitor oxygen levels. A probe placed on the hand or foot can be used to monitor oxygen levels all the time (continuous oxygen monitoring) or just every 4-6 hours (intermittent oxygen monitoring). Research has suggested that placing infants with bronchiolitis on continuous monitoring results in unnecessary use of oxygen and infants staying longer in hospital. However, due to the lack of high quality research, its unclear which strategy is best and practice varies. The objective of this study is to conduct high quality research across hospitals to determine whether intermittent compared to continuous oxygen monitoring will reduce the length of hospital stay in infants hospitalized with bronchiolitis. The investigators will also compare safety and cost. The results of this study will inform bronchiolitis practice standards and the best use of health care resources.

DETAILED DESCRIPTION:
BACKGROUND This research protocol focuses on bronchiolitis, a leading cause of infant hospitalization and cumulative expense for the health care system. Supportive management, such as oxygen supplementation and monitoring, is the major focus of care, as active medical treatment is not effective. Oxygen saturation monitoring may be performed on an intermittent (e.g. every 4-6hrs) or continuous basis for stable infants hospitalized with bronchiolitis. Observational studies find that the use of continuous monitoring is associated with overuse of supplemental oxygen and longer hospital stay. Based on this low quality evidence, practice guidelines state that clinicians may choose not to use continuous monitoring and practice variation exists due to a lack of RCTs.

SPECIFIC AIMS Primary: To determine if intermittent vs continuous oxygen saturation monitoring will reduce length of hospital stay in infants with bronchiolitis. Secondary: To determine differences in other outcomes - effectiveness, safety, acceptability, and cost.

METHODOLOGY Design: multi-centre, pragmatic, parallel group, 1:1, two arm superiority RCT. Population: Previously healthy infants (4 weeks-2 years) hospitalized with bronchiolitis who are clinically stable, will be recruited from children's and community hospitals in Ontario, Canada.

Interventions: Randomization to intermittent (every 4hrs) or continuous oxygen saturation monitoring. In keeping with local and national clinical practice guidelines, an acceptable oxygen saturation target of ≥ 90% will be used for both groups.

ELIGIBILITY:
Children admitted to the general pediatric inpatient unit (GPIU) with bronchiolitis will be eligible if their clinical status is stable and not at high risk of deterioration

Inclusion Criteria:

* Clinical diagnosis of bronchiolitis as determined by the attending physician.
* First episode of acute bronchiolitis.
* Age: 4 weeks to 24 months.
* Clinical status stable for 6 hours
* Parent consent

Exclusion Criteria:

* Known risk factors for clinical deterioration including chronic medical condition; premature birth (<35weeks), history of apnea, weight < 4kg, receiving morphine
* Patient on heated high flow oxygen at enrolment
* ICU admission on current admission
* No telephone available

Ages: 4 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay from randomization on the inpatient unit to discharge from hospital | 1 month

SECONDARY OUTCOMES:
Duration of oxygen supplementation from randomization to discontinuation of supplementation | 1 month
Number of medical interventions performed from time of randomization to hospital discharge | 1 month
Time from randomization to meeting hospital discharge criteria | 1 month
Length of hospital stay from inpatient unit admission to hospital discharge | 1 month
Parent anxiety | 1 month
  Parents will rate their level of anxiety at the current time (state anxiety) and generally (trait anxiety) from the adult State Trait Anxiety Inventory questionnaire during the hospital stay.
Number of parent work days missed from randomization to 15 days after discharge | 15 days after discharge
Nursing satisfaction | 1 month
  The attending nurse will be asked to complete a 10 mm visual analogue scale (VAS) to measure their satisfaction with the quality of monitoring.
PICU admission after randomization | 1 month
PICU consultation after admission | 1 month
Unscheduled return to care within 15 days of discharge | 15 days after discharge
Mortality | 15 days after discharge.
Cost-Effectiveness | 15 days after discharge.
  Cost-effectiveness will be measured by the incremental cost-effectiveness ratio (ICER), a ratio defined by the incremental difference in costs between treatment arms and the incremental difference in length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Mahant, Principal Investigator — The Hospital for Sick Children
Locations (6):
- Canada (6):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Trillium Health Partners (Credit Valley Site), Mississauga, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahant S, Wahi G, Bayliss A, Giglia L, Kanani R, Pound CM, Sakran M, Kozlowski N, Breen-Reid K, Arafeh D, Moretti ME, Agarwal A, Barrowman N, Willan AR, Schuh S, Parkin PC; Canadian Paediatric Inpatient Research Network (PIRN). Intermittent vs Continuous Pulse Oximetry in Hospitalized Infants With Stabilized Bronchiolitis: A Randomized Clinical Trial. JAMA Pediatr. 2021 May 1;175(5):466-474. doi: 10.1001/jamapediatrics.2020.6141. PMID 33646286
- [Derived] Mahant S, Wahi G, Giglia L, Pound C, Kanani R, Bayliss A, Roy M, Sakran M, Kozlowski N, Breen-Reid K, Lavigne M, Premji L, Moretti ME, Willan AR, Schuh S, Parkin PC. Intermittent versus continuous oxygen saturation monitoring for infants hospitalised with bronchiolitis: study protocol for a pragmatic randomised controlled trial. BMJ Open. 2018 Apr 20;8(4):e022707. doi: 10.1136/bmjopen-2018-022707. PMID 29678995